CLINICAL TRIAL: NCT01275911
Title: Fast-track Laparoscopic Surgery. The Effect of Anesthetic Technique
Brief Title: Non-opioid Analgesia for Fast-track Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Gabriele Baldini, MD, MSc, Assistant Professor, MD, MSc, Anesthesiologist, Assistant Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GEN#08-22
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Last update posted 2013-03-27 (Estimated); Status verified 2013-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — esmolol; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Esmolol (Experimental)
  Interventions: Drug: Esmolol
- Remifentanil (Active Comparator)
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Esmolol — Induction of anesthesia: 1mg/Kg; Maintenance during surgery: 5-15 mcg/kg/min
  Arms: Esmolol
Drug: Remifentanil — At the induction of anesthesia: 1mcg/Kg; Maintenance during surgery: 0.025-0.25mcg/kg/min
  Arms: Remifentanil

SUMMARY:
In this randomized observer-blinded trial the analgesic efficacy of intravenous esmolol, as alternative to intraoperative opioids, is tested in patients undergoing laparoscopic prostatectomy and upper gastrointestinal surgery (such as Nissen fundoplication). The purpose of this study is to determine whether intravenous esmolol improves postoperative analgesia and accelerate the surgical recovery. We hypothesize that patients receiving intravenous esmolol will consume less analgesic in the postoperative period, will have less opioid-related side effects and will recover their functional status faster then patients receiving intravenous esmolol.

Patients will be stratified according to the type of surgical procedure in 2 arms: 40 patients with prostate cancer and undergoing elective laparoscopic prostatectomy, and 40 patients with gastro-esophageal reflux undergoing upper gastrointestinal surgery (Nissen funduplication) will be enrolled.

Patients will receive total intravenous anesthesia with propofol and esmolol (Esmolol group, n=20 in each arm) or propofol and remifentanil (Remifentanil Group, n=20 in each arm).

DETAILED DESCRIPTION:
Outcomes:

1. Primary: The amount of fentanyl needed in PACU and the amount of PCA morphine used during the first 24 postoperative hours.
2. Secondary: intensity of postoperative pain (visual analogue scale,VAS), opioids side effects, length of stay in PACU and in the hospital, short-term SF-36 questionnaire, CHAMPS questionnaire, and the 2 and 6 minutes walking tests.

Methodology:

In each arm patients will be assigned by computer generated random letters to two groups:

The Esmolol group: patients will receive no opioids but will receive esmolol at induction and as a continuous infusion during the surgery.

The Remifentanil group: patients will receive remifentanil as sole opioid during induction of anesthesia as a continuous infusion during the surgery.

During the preoperative assessment patients will be asked to fill out the CHAMPS and the Short-term SF-36 questionnaires. The 2 and 6 minutes walking tests will be also administered

On arrival in the operating room, routine monitors will be applied for recording heart rate, systolic blood pressure, and oxygen saturation. In addition, the electroencephalographic bispectral index (BIS) value was obtained using a single channel sensor in a frontal temporal area. The BIS is a standard monitor of depth of anesthesia and measures cortical activation. It has been found to be well correlated to electroencephalogram. After obtaining baseline values, midazolam 1-2mg IV will be administered for pre-medication. Anesthesia will be subsequently induced with Propofol 2-2.5 mg/kg, Rocuronium 0.45-0.9 mg/kg.

The Esmolol group will receive 1.0 mg/kg of esmolol and the Remifentanil group 1.0 mcg/kg of remifentanil for induction of anesthesia. After direct laryngoscopy and tracheal intubation will have been performed, anesthesia will be maintained with a continuous infusion of propofol 80-250 mcg/kg/min to maintain a "targeted" BIS value of 50 or less (BIS below 60 signifies the patient is asleep and unaware, 90 and over signifies intraoperative wakefulness). Patients will receive either esmolol infusion of 5-15 mcg/kg/min or remifentanil infusion of 0.025-0.25mcg/kg/min (in Esmolol group or in the Remifentanil group respectively) titrated to maintain HR within 25% of the pre-induction baseline value with targeted HR in between 55-90. Furthermore, the patients will also receive IV fluid at 6 ml/kg. All patients will be mechanically ventilated to maintain the end-tidal carbon dioxide (CO2) concentration in the range of 36-44 mm Hg and will receive toward the end of surgery Ketorolac 30mg IV, Droperidol 0.625mg IV and neuromuscular reversal if needed. Propofol will be discontinued after the last skin suture and the remifentanil or esmolol infusions will be stopped. After closure 10cc of bupivacaine 0.25% with epinephrine 1:200.000 will be infiltrated in the surgical ports. Nurses in the PACU will be informed that patients are taking part of the study but will not be aware of the hypothesis and will provide patients with standard care. Patients will have access in PACU to Fentanyl 25mcg IV q5min and to Ondansetron 2-8mg IV prn (standard medications used in this institution). Patients will receive PCA morphine for 24-48 h with tylenol 650mg PO q4h and naproxen 500mg or celebrex 200 mg PO bid.

Heart rate, blood pressure, BIS and oxygen saturation will be recorded at baseline, induction of anesthesia, tracheal intubation, skin incision, and subsequently at 5 min intervals until the end of surgery. Patients will be extubated in the operating room. They will then be transported to the post anesthesia care unit (PACU).

Assessment:

Recovery time will be assessed by a blinded observer (research fellow) unaware of the study hypothesis from the time the study drugs are discontinued. Times to awakening (opening eyes on verbal command), and orientation to person, date and place will be recorded, whereas the time to home readiness will be evaluated using standardized discharge criteria as described by White-Song17 at 30 min intervals. The score maximum of 12 out of 14 allows the patients to be discharged to the surgical ward from the PACU. Pain will be assessed every 15 minutes using (visual analog scale) (VAS)18 (0-10 cm) at rest, on movements and on coughing by the recovery nurse. Postoperative side effects (nausea, vomiting, pain), requirement for analgesics and antiemetics therapy (morphine and zofran respectively), as well as patient satisfaction will be assessed on discharge from PACU and 24-48 hrs after the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with prostate cancer undergoing laparoscopic prostatectomy
2. Patients with gastro-esophageal reflux undergoing upper abdominal surgery (Nissen funduplication)

Exclusion Criteria:

1. Age <18 yr or > 85 yr
2. ASA physical status 3 and greater
3. History of hepatic failure (Child & Pug A-C)
4. Renal failure (creatinine outside the normal range)
5. Cardiac failure (NYHA I-IV)
6. Organ transplant
7. Diabetes mellitus type 1 and 2
8. Morbid obesity (BMI > 40)
9. Chronic use of opioids and beta-blockers
10. Severe mental impairment
11. History of allergic reactions to all the medications used in the study or inability to understand pain assessment.
12. Asthma or Reactive airway disease
13. Patient with known or suspected peritoneal adhesion
14. Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-01; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Amount of postoperative opioid consumption | End of surgery- 24hr from the end of surgery

SECONDARY OUTCOMES:
Postoperative pain intensity | every 24 hr from the end of surgery
Incidence of opioids side-effects | during the duration of hospital stay
Length of stay in the PACU | time spent in the recovery room
Length of stay in the hospital | duration of hospitalization after the surgery
CHAMPS questionnaire | preoperative, at 3 and 8 weeks after the surgery
short-term SF-36 | preoperative, at 3 and 8 weeks after the surgery
2 minutes walking test | preoperative, at 4 weeks after the surgery
6 minutes walking test | preoperative, at 4 weeks after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Baldini, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Montreal General Hospital, McGill University Health Centre, Montreal, Quebec, Canada

REFERENCES:
- [Result] Collard V, Mistraletti G, Taqi A, Asenjo JF, Feldman LS, Fried GM, Carli F. Intraoperative esmolol infusion in the absence of opioids spares postoperative fentanyl in patients undergoing ambulatory laparoscopic cholecystectomy. Anesth Analg. 2007 Nov;105(5):1255-62, table of contents. doi: 10.1213/01.ane.0000282822.07437.02. PMID 17959952
- [Result] Coloma M, Chiu JW, White PF, Armbruster SC. The use of esmolol as an alternative to remifentanil during desflurane anesthesia for fast-track outpatient gynecologic laparoscopic surgery. Anesth Analg. 2001 Feb;92(2):352-7. doi: 10.1097/00000539-200102000-00014. PMID 11159231
- [Result] Johansen JW, Schneider G, Windsor AM, Sebel PS. Esmolol potentiates reduction of minimum alveolar isoflurane concentration by alfentanil. Anesth Analg. 1998 Sep;87(3):671-6. doi: 10.1097/00000539-199809000-00034. PMID 9728851
- [Result] White PF, Wang B, Tang J, Wender RH, Naruse R, Sloninsky A. The effect of intraoperative use of esmolol and nicardipine on recovery after ambulatory surgery. Anesth Analg. 2003 Dec;97(6):1633-1638. doi: 10.1213/01.ANE.0000085296.07006.BA. PMID 14633533
- [Result] Chia YY, Chan MH, Ko NH, Liu K. Role of beta-blockade in anaesthesia and postoperative pain management after hysterectomy. Br J Anaesth. 2004 Dec;93(6):799-805. doi: 10.1093/bja/aeh268. Epub 2004 Sep 17. PMID 15377583
- [Result] Erdil F, Demirbilek S, Begec Z, Ozturk E, But A, Ozcan Ersoy M. The effect of esmolol on the QTc interval during induction of anaesthesia in patients with coronary artery disease. Anaesthesia. 2009 Mar;64(3):246-50. doi: 10.1111/j.1365-2044.2008.05754.x. PMID 19302635
- [Result] Smith I, Van Hemelrijck J, White PF. Efficacy of esmolol versus alfentanil as a supplement to propofol-nitrous oxide anesthesia. Anesth Analg. 1991 Nov;73(5):540-6. PMID 1683182
- [Result] White PF. The role of non-opioid analgesic techniques in the management of pain after ambulatory surgery. Anesth Analg. 2002 Mar;94(3):577-85. doi: 10.1097/00000539-200203000-00019. No abstract available. PMID 11867379